CLINICAL TRIAL: NCT06366815
Title: Characterizing Phenothypes in Non Ambulant Duchenne Muscular Dystrophy
Brief Title: phenotypeS in Non Ambulant Duchenne Muscular Dystrophy
Acronym: GUP21003
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Pane Marika, prof associate, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4619
Record Dates: First submitted 2023-02-08; First posted 2024-04-16 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Duchenne Muscular Dystrophy; Natural History; Motor Function; Retardation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Different Phenotypes of non ambulant patients with Duchenne Muscular Dystrophy — clinical and functional data collection of non ambulant patients with Duchenne muscular dystrophy

SUMMARY:
The aims of the study are to prospectively collect information on several aspects of function in non-ambulant DMD patients by using a structured battery of tests including motor, respiratory and cardiac function

DETAILED DESCRIPTION:
The aims of the study are to prospectively collect information on several aspects of function in non-ambulant DMD patients by using a structured battery of tests including motor, respiratory and cardiac function, to retrospectively review similar information on the data collected in the last decade and to establish the effect of steroids after loss of ambulation on different aspects of function.

We also aim to use this integrated approach to identify patterns of severity and progression, the most appropriate outcome measures and endpoints in each group and possible genotype/phenotype correlations.

ELIGIBILITY:
Inclusion Criteria:

* Children with genetically confirmed diagnosis of Duchenne Muscular Dystrophy will be included in the study. We will include all Duchenne Muscular Dystrophy boys who have lost the ability to walk independently.
* All patients in whom consent can be obtained will be enrolled with no exclusion criteria.

Exclusion Criteria:

* Patients lacking genetic confirmation of Duchenne Muscular Dystrophy
* Patients still able to walk for more than 10 meters.

Ages: 8 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Population expected to be enrolled will include almost 250 patients affected from Duchenne Muscular Dystrophy with a confirmed genetic diagnosis and that have lost the ability to walk indipendently for more than 10 meters.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
motor function | 24 months
  assessment of Upper Limb Motor function in all the patient at baseline, 6, 12 and 24 months
respiratory function | 24 months
  Assessment of respiratory function, in particular Forced Vital Capacity at baseline, 6, 12 and 24 months in all the patients able to perform the test. Registration of need for ventilation and hours of ventilation needed at each assessment
cardiac function | 24 months
  Assessment of ejection fraction through cardiac ultrasound at baseline and changes at follow up assessment at 6, 12 and 24 months

SECONDARY OUTCOMES:
identify patterns of severity and of progression related to differnt genotypes | 24 months
  evaluation correlation genotype/phenotype

CONTACTS AND LOCATIONS:
Overall Officials: Marika Pane, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (2):
- Italy (2):
  - IRCCS Eugenio Medea - Ass. "La Nostra Famiglia", Bosisio Parini, Lc
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: No